CLINICAL TRIAL: NCT03443648
Title: Fixator Assisted Plating for Correction of High Degree Genu Varum Deformity
Brief Title: External Fixator Assisted Genu Varum Correction
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Kerolos Maged, Resident in the orhtopaedics and traumatology department, Assiut University
Allocation: Not Applicable | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: FAVC
Record Dates: First submitted 2017-11-25; First posted 2018-02-23 (Actual); Last update posted 2018-05-01 (Actual); Status verified 2018-04

CONDITIONS: Deformity
MeSH Terms: conditions — Congenital Abnormalities

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: External fixator assisted plaing — The plate length is marked on the skin. Limb reconstruction system (LRS) with one swivel clamp or Taylor Spatial frame (TSF) is used in all cases. The fixator is put in a plane parallel to that of the deformity. Two tapered pins are placed on either side of the planned osteotomy site and passed at a distance from the osteotomy so that they will not impede the subsequent internal fixation. Swivel clamps or the struts of the TSF are aligned in such a way that full correction is achieved. After osteotomy, swivel clamp is loosened and angular correction is achieved. Translation is carried out according to preoperative planning. If readjustment is required the swivel clamps or TSF struts are loosened and further correction is carried out. Once desired correction is achieved, the clamps or struts are tightened. Definitive internal fixation is carried out while external fixation holds the fragments. For internal fixation, locked T plate will be used.

SUMMARY:
Assessment of accuracy of correction of genu varum more than 20 degrees using external fixator assisted plating. Intraoperatively, the operative time needed for completion of accurate correction, torniquet use, blood loss will be assessed. Postoperative complications either early ones like infection, thromboembolic complications, peroneal nerve palsy or late post operative complications like implant failure, delayed union, non union and bone healing time will be assessed..

DETAILED DESCRIPTION:
Malalignment prevents proper transmission of forces across the knee leading to advance or even start the progression of osteoarthritis.Preoperative planning is necessary to identify the level and magnitude of the deformity. Corrections can be performed acutely or gradually. Acute correction can be achieved by opening wedge, closing wedge or dome osteotomies followed by internal fixation. On the other hand, gradual correction can be achieved by osteotomy with external fixation.

Although osteotomy with internal fixation is more convenient to the patient than external fixator, it has many drawbacks. These include the need for large surgical exposure, soft tissue stripping and difficulty executing precise deformity correction. Meticulous preoperative planning is important when internal fixation is planed. It also needs to be executed precisely till fixation is completed. Under-correction or over-correction is possible while executing the procedure. Furthermore, iatrogenic deformity in other planes may also develop. If such a deformity is significant, it may adversely affect the function or may lead to excessive loading on adjacent joints. In some cases, revision of surgery for further correction may be required to correct this residual or iatrogenic deformity.

External fixation can be used for gradual correction of genu varum. In spite of the disadvantages of external fixation like being uncomfortable for the patient, tethering soft tissue, associated pin site infection and irritation , it is re-adjustable postoperatively. This allows controlled accurate correction of the mechanical axis of the lower limb.

Our study is implicated on correction of high degree genu varum which is more than 20 degrees .To correct such deformity, it is difficult to calculate the amount of wedge opening intraoperative. The described trigonometric calculation of the size of the base is described for deformity less than 20 degrees .In this study we are going to use a hybrid technique of both external and internal fixation, so we can make use of the benefits of both internal and external fixation techniques External fixation by limb reconstruction system (LRS) or Taylor Spatial frame(TSF) is used to control and stabilize fragments while performing the desired correction. A locked T plate is then applied to stabilize the fully corrected osteotomy. This allows intraoperative removal of the external fixator without loss of correction. Then we compare the planned correction with the achieved correction.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18years old or more
2. Varus 20 degrees or more

Exclusion Criteria:

1. Contraindication to internal fixation
2. Associated osteoarthritis

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Estimated)
Dates: Start 2018-06-01 (Estimated); Primary Completion 2020-03-31 (Estimated); Study Completion 2020-03-31 (Estimated)

PRIMARY OUTCOMES:
assesment of accuracy of correction of high degree genu varum using this method of correction. | one year
  assessment of mechanical axis deviation in degrees, mechanical tibiofemral angle in degrees, medial proximal tibial angle in degrees and the position of mechanical axis ratio. They are all measured in the immediate post operative long film and the long film after one year. The normal angles are known documented angles so, we will compare the preoperative and postoperative angles with the normal ones.Immediate postoperative long film on the lower limbs to compare pre and postoperative angles with the normal angles. Another long film is done after one year to follow up the achieved correction

REFERENCES:
- [Background] Hochberg MC, Altman RD, Brandt KD, Clark BM, Dieppe PA, Griffin MR, Moskowitz RW, Schnitzer TJ. Guidelines for the medical management of osteoarthritis. Part II. Osteoarthritis of the knee. American College of Rheumatology. Arthritis Rheum. 1995 Nov;38(11):1541-6. doi: 10.1002/art.1780381104. PMID 7488273
- [Background] Sharma L, Song J, Felson DT, Cahue S, Shamiyeh E, Dunlop DD. The role of knee alignment in disease progression and functional decline in knee osteoarthritis. JAMA. 2001 Jul 11;286(2):188-95. doi: 10.1001/jama.286.2.188. PMID 11448282
- [Background] Hernigou P, Medevielle D, Debeyre J, Goutallier D. Proximal tibial osteotomy for osteoarthritis with varus deformity. A ten to thirteen-year follow-up study. J Bone Joint Surg Am. 1987 Mar;69(3):332-54. PMID 3818700
- [Background] Tuli SM, Kapoor V. High tibial closing wedge osteotomy for medial compartment osteoarthrosis of knee. Indian J Orthop. 2008 Jan;42(1):73-7. doi: 10.4103/0019-5413.38585. PMID 19823659
- [Background] Sundaram NA, Hallett JP, Sullivan MF. Dome osteotomy of the tibia for osteoarthritis of the knee. J Bone Joint Surg Br. 1986 Nov;68(5):782-6. doi: 10.1302/0301-620X.68B5.3782246.
- [Background] Rozbruch SR, Segal K, Ilizarov S, Fragomen AT, Ilizarov G. Does the Taylor Spatial Frame accurately correct tibial deformities? Clin Orthop Relat Res. 2010 May;468(5):1352-61. doi: 10.1007/s11999-009-1161-7. Epub 2009 Nov 13. PMID 19911244
- [Background] Kazemi SM, Qoreishi M, Behboudi E, Manafi A, Kazemi SK. Evaluation of Changes in the Tibiotalar joint after High Tibial Osteotomy. Arch Bone Jt Surg. 2017 May;5(3):149-152. PMID 28656162
- [Background] Gugenheim JJ Jr, Brinker MR. Bone realignment with use of temporary external fixation for distal femoral valgus and varus deformities. J Bone Joint Surg Am. 2003 Jul;85(7):1229-37. doi: 10.2106/00004623-200307000-00008. PMID 12851347
- [Background] Bar-On E, Becker T, Katz K, Velkes S, Salai M, Weigl DM. Corrective lower limb osteotomies in children using temporary external fixation and percutaneous locking plates. J Child Orthop. 2009 Apr;3(2):137-43. doi: 10.1007/s11832-009-0165-x. Epub 2009 Mar 12. PMID 19308625
- [Background] Rozbruch SR. Fixator-assisted plating of limb deformities. Oper Tech Orthop. 2011;21:174-.
- [Background] Insall JN, Dorr LD, Scott RD, Scott WN. Rationale of the Knee Society clinical rating system. Clin Orthop Relat Res. 1989 Nov;(248):13-4. PMID 2805470
- [Background] Tegner Y, Lysholm J. Rating systems in the evaluation of knee ligament injuries. Clin Orthop Relat Res. 1985 Sep;(198):43-9. PMID 4028566
- [Background] Paley D, Herzenberg JE, Tetsworth K, McKie J, Bhave A. Deformity planning for frontal and sagittal plane corrective osteotomies. Orthop Clin North Am. 1994 Jul;25(3):425-65. PMID 8028886
- [Background] Paley D. 1st ed. New York: Springer; 2002. Principles of deformity correction; p 1-18.12.
- [Background] Paley D. 1st ed. New York: Springer; 2002. Principles of deformity correction; pp. 175-94